CLINICAL TRIAL: NCT07078162
Title: Accuracy Of Fitting Surface Of Orbital Prosthesis Constructed By Photogrammetry Scan
Acronym: OrbitalProsth
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tanta University (Other)
Responsible Party: Principal Investigator, Asmaa Abd Allah Hassan Hashish, Principal Investigator (Teaching Assistant in Prosthdontic Department), Tanta University
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: Orbital prosthesis; 2950729 (Other: faculty of dentistry - Tanta University)
Record Dates: First submitted 2025-07-01; First posted 2025-07-22 (Actual); Last update posted 2025-07-22 (Actual); Status verified 2025-06

CONDITIONS: Orbital Deformity
Keywords: Orbital Prosthesis; Photogrammetry; Impression; 3D printing; Silicone; Accuracy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 1- photogrammetry scan to the defect and healthy sites (Other): Capture photographs of the face including the defective site by profesional camera
  Interventions: Other: Photogramety Orbital Prosthesis
- 2- Digital scan of a conventional impression to the defect and healthy sites (Other): Digital scan of a conventional impression to the defect and healthy sites, the impression was taken using silicone rubber impression material, to obtain 3D virtual model using an extraoral desktop scanner.
  Interventions: Other: Conventional impression prosthesis

INTERVENTIONS:
Other: Photogramety Orbital Prosthesis — Using 2D photographs to abtain 3D model of orbital defect anatomy
  Arms: 1- photogrammetry scan to the defect and healthy sites
Other: Conventional impression prosthesis — Conventional impression to an orbital defect then scaning the impression using desktop scanner
  Arms: 2- Digital scan of a conventional impression to the defect and healthy sites

SUMMARY:
Two orbital prosthesis were made to the patient , using two different digital scanning methods to restore the unilateral orbital exentration , the prosthetic devices were made using medical silicon material

DETAILED DESCRIPTION:
Statement of problem : Orbital defects which resulted from surgical removal of mucormycosis that caused by corona virus infection lead to several functional, esthetic and psychological problems for the patients.

Aim of the study : Evaluation of the accuracy of fitting surface of orbital prosthesis constructed by photogrammetry scan.

Methods : An orbital prosthesis was made using photogrammetry scanning technique as a method for making digital facial impression to obtain facial 3D model using a high resolution professional camera with image processed through 3DF Zephyr open-source software and the other orbital prosthesis was made using a conventional impression for both the defect and contralateral healthy eye , then scanned with a Degree Of Freedom (DOF) extra oral desktop scanner. 3D models of the defect sites were printed from each scanning method to act as a master cast for the orbital prosthesis fabrication. Accuracy of orbital prosthesis fitting surfaces produced from the two techniques in comparison with a facial scan as a reference scan was assessed through deviation analysis using metrology grade software (Geomagic Control X ).

ELIGIBILITY:
Inclusion Criteria:

1. Patients with Unilateral orbital defect.
2. Complete healing of the defect site with no open wound.
3. At least 1 year passed after the last chemo or radiotherapy dose in patients who receiving this type of treatment

Exclusion Criteria:

1. Patient under chemo or radiotherapy due to presence of active tumor.
2. Patient with unhealed

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2024-06-23 (Actual); Primary Completion 2025-04-23 (Actual); Study Completion 2025-06-23 (Actual)

PRIMARY OUTCOMES:
Accuracy of fitting surface of orbital prosthesis | Baseline or Day 1
  Measurements of accuracy:
  Measuring surfaces mesh deviation between the two orbital prosthesis fitting surfaces obtained using two types of scanning methods and a reference facial scan obtained using creality raptor (CR) scanner.
  1. The STL file of the facial scan and the STL files of the two orbital prosthesis fitting surfaces were imported separately to the metrology grade software program( Geomagic control x) .
  2. The STL file of the facial scan was selected and considered to be the reference data , and the STL files of the prosthesis fitting surfaces was selected and considered to be the measured data .
  3. The STL file of the measured data was manually superimposed onto the STL file of the reference data .
  4. A color surface map appeared on the reference data which indicate the directional mesh deviation result between the superimposed scans .
  5. The color map scale was adjusted .

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Dentistry Tanta University, Tanta, Egypt

IPD SHARING:
Plan to Share IPD: No
for the patient privacy